CLINICAL TRIAL: NCT03343873
Title: The Effects of Different Anesthetics on Functional Connectivity in Volunteers and Patients With Brain Tumor (ACTION)
Brief Title: The Effects of Different Anesthetics on Functional Connectivity
Acronym: ACTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2017-7-17
Record Dates: First submitted 2017-09-17; First posted 2017-11-17 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Sedation
Keywords: anesthetics; fMRI; functional connectivity
MeSH Terms: interventions — Midazolam; Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Midarolam (Experimental): midarolam sensation group
  Interventions: Drug: Midazolam
- Propofol (Experimental): propofol sensation group
  Interventions: Drug: Propofol
- dexmedetomidine (Experimental): dexmedetomidine sensation group
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — Midazolam was administered intravenously at a dose of 0.1 mg / kg followed by continuous intravenous injection at 0.03 mg / kg / h and maintained until the course of the scan.
  Arms: Midarolam
Drug: Propofol — Propofol group 1mg / kg intravenous injection, followed by 2mg / kg / h continuous intravenous injection, and maintained to the scanning process;
  Arms: Propofol
Drug: Dexmedetomidine — Dexmedetomidine group with total amount of 1μg / kg, infusion time 15min, followed by 0.6μg / kg / h, and maintained to the scanning process;
  Arms: dexmedetomidine

SUMMARY:
This research is a prospective cohort study. The aim of the study is to determine different levels of sedative mechanism and the effect on brain functional connectivity of midazolam, dexmedetomidine and propofol.

DETAILED DESCRIPTION:
This research will include 120 healthy volunteers and 120 brain tumor patients; the participants will be allocated into midazolam, dexmedetomidine and propofol group. Resting and task fMRI will be performed at awake (BIS>90), mild sedation (BIS 80-85), moderate sedation (BIS 65-75), deep sedation (BIS 45-55) and recovery states (BIS >90). The primary outcome of our study is the effect of different levels of sedation for brain network connection. The secondary outcomes are the effect of different levels of sedation for default, executive control, sensory and motor networks and their subnetwork connectivity; the sedation state, circulatory and respiratory parameters of the participants, and the adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male, 18 ~ 65 years old
* 2. Healthy Volunteer / Brain Tumor Patients
* 3. Senior high school and above
* 4. Sign informed consent

Exclusion Criteria:

* 1. In vivo implant MRI check taboo
* 2. Cardiopulmonary liver and kidney and other systemic complications
* 3. History of major surgical anesthesia
* 4. Abuse of drugs, alcoholism history
* 5. Test drug allergy history
* 6. Claustrophobia
* 7. Left hand

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude of Low Frequency Fluctuations（ALLF）and Regional Homogeneity（ReHo) | 30mins after administration
  The differences of amplitude of low frequency fluctuations (ALFF/Low Frequency Amplitude) and regional homogeneity（ReHo) in brain voxel - wise under anesthetic sedations.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph.D, Study Chair — Department of Anesthesiology, Beijing Tiantan Hospital
Locations (1):
- Beijing Tian Tan Hospital, Beijing, China